CLINICAL TRIAL: NCT02359851
Title: A Multicenter Phase II Study to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) in Patients With Advanced Uveal Melanoma
Brief Title: Pembrolizumab in Treating Patients With Advanced Uveal Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Douglas Johnson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC MEL1486; NCI-2015-00020 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2015-02-04; First posted 2015-02-10 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Stage IIIA Uveal Melanoma; Stage IIIB Uveal Melanoma; Stage IIIC Uveal Melanoma; Stage IV Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with uveal melanoma that has spread to other places in the body and usually cannot be cured or controlled with treatment. Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate objective response rate (ORR) in patients with advanced uveal melanoma receiving pembrolizumab.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) in patients with advanced uveal melanoma receiving pembrolizumab.

II. To evaluate safety, tolerability and adverse experience profile of pembrolizumab in uveal melanoma.

III. To evaluate overall survival (OS) in patients with advanced uveal melanoma receiving pembrolizumab.

TERTIARY OBJECTIVES:

I. To evaluate objective response rate (ORR; complete response + partial response) in patients with advanced uveal melanoma receiving pembrolizumab as stratified by programmed cell death-ligand 1 (PD-L1) expression and guanine nucleotide-binding protein (GNA)Q/GNA11 mutation status.

II. To evaluate ORR in patients previously treated with ipilimumab or with mitogen-activated protein kinase kinase (MEK) inhibitors.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Histologic confirmation of advanced (metastatic or unresectable) uveal melanoma. If uveal melanoma has been diagnosed clinically and/or by gene expression profiling, patients may be included following discussion with the principal investigator.
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN; creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-cluster of differentiation (CD)137; patients who received anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) (ipilimumab, tremelimumab) will NOT be excluded and are eligible for inclusion
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnson, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Johnson DB, Bao R, Ancell KK, Daniels AB, Wallace D, Sosman JA, Luke JJ. Response to Anti-PD-1 in Uveal Melanoma Without High-Volume Liver Metastasis. J Natl Compr Canc Netw. 2019 Feb;17(2):114-117. doi: 10.6004/jnccn.2018.7070. PMID 30787124
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this trial was May 2015 to January 2017. The trial was conducted at Vanderbilt-Ingram Cancer Center in Nashville, Tennessee and University of Chicago in Chicago, Illinois This trial closed due to slow accrual.
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 5
Completed | 3
Not Completed | 2
Not completed — Death | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (16.7332)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Defined as the Percentage of Patients Achieving a Confirmed Complete or Partial Response, as Defined by Immune-related Response Criteria (irRC)
Description: Of note, response rates by RECIST 1.1 criteria will also be assessed although irRC will be used for the primary endpoint. The percentage of complete or partial response is calculated and 95% confidence interval is estimated using Wilson method.
Time Frame: Up to 3 years
Population: Patients received pembrolizumab treatment and evaluated for response.
Measure: Mean (95% Confidence Interval); unit: % of patients achieving response
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 4
% of patients achieving response | 25 [1.3 to 69.9]

2. Secondary Outcome: Progression-Free Survival (PFS) Defined as Time From Treatment to Progression Defined by RECIST1.1 Criteria or Death.
Description: PFS will be summarized using the method of Kaplan and Meier. Median PFS time with 95% confidence intervals will be reported. Using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), progression will be defined as ≥ 20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest diameter recorded or the appearance of one or more new lesions, and/or appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions.
Time Frame: Time from the first dose of pembrolizumab to progression, assessed up to 3 years.
Population: Patients received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 5
months | 36.0 [NA to NA] — Insufficient patient data.

3. Secondary Outcome: Overall Survival (OS) Defined as Number of Patients Surviving up to 3 Years.
Description: The Kaplan-Meier method will be used to estimate the overall survival. Median survival and its 95% confidence interval will be estimated and reported.
Time Frame: Interval between the first dose of pembrolizumab and death for any reason, assessed up to 3 years
Population: Patients received pembrolizumab treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 5
Participants
  Survived | 3
  Died | 2

4. Secondary Outcome: Response Duration
Description: If sample size permits, response duration will be summarized descriptively using Kaplan-Meier medians and quartiles. Only the subset of patients who show a complete response or partial response will be included in this analysis.
Time Frame: Up to 3 years
Population: Only 1 participant had a RECIST-defined response, which is ongoing and lasting 23.5 months.
Measure: Number; unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 1
months | 23.5

5. Secondary Outcome: Number of Patients With Each Worst-Grade Toxicity. Incidence of Adverse Events, Using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening; grade 5, death. This endpoint will be reported descriptively without formal statistical analysis.
Time Frame: Up to 30 days after the last dose of trial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 4
Participants
  Number of participants with worst-grade toxicity 1 | 1
  Number of participants with worst-grade toxicity 2 | 1
  Number of participants with worst-grade toxicity 3 | 0
  Number of participants with worst-grade toxicity 4 | 1
  Number of participants with worst-grade toxicity 5 | 1

6. Other Pre Specified Outcome: Changes in GNAQ/GNA11 Mutation Status on Each Patient Per Institutional Protocol
Description: Differences in PFS and OS between subgroups will be assessed by the stratified logrank test. Differences in ORR between subgroups will be assessed by the Pearson chi-square test. No adjustments will be made for multiple comparisons.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in PD-L1 Expression Status on Archival or Fresh Tissue From All Patients and Correlate With ORR
Description: as for outcome 6
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Molecular Characteristics of Uveal Melanoma When Treated With Pembrolizumab
Description: Each relevant clinical characteristic will be recorded by the use of tables and/or graphs. The number and percentage of patients treated, and the primary reason for discontinuation will be displayed. Demographic variables (such as age) and baseline characteristics will be summarized by descriptive statistics. Compliance with pembrolizumab administration will be measured by patients: 1) receiving unscheduled study agent infusions/injections; 2) missing an infusion/injection. Numbers and percentages of patients and infusion/injection visits with any deviation in these measures will be reported.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time participants signed consent form through 30 days following cessation of treatment .
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=5)
Increased Creatinine (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
INR Increased (Investigations) | 1 (1)
Acute Kidney Inury (Renal and urinary disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lower GI Hemorrhage (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Perforate diverticulitis (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Neoplassms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=5)
Fatigue (General disorders) | 3 (5)
Limb edema (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (7)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (5)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dry Eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Retinal vascular disorder (Eye disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02359851/Prot_SAP_000.pdf